CLINICAL TRIAL: NCT01027624
Title: Centralized Pan-South African Survey on the Undertreatment of Hypercholesterolaemia.
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Pharmaceuticals Pty Ltd
Other Study IDs: NIS-CZA-DUM-2009/1
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Undertreatment of Hypercholesterolaemia
Keywords: Pan South African Survey on the Undertreatment of Hypercholesterolaemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hyperchlesterolaemia: Participants undertreated with hypercholesterolaemia

SUMMARY:
This is a multi-centre survey of patients who are currently on lipid lowering pharmacological treatment in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older of either gender or race.
* Subject must provide informed consent and comply with the survey procedures.
* Subject is on lipid lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-centre survey of patients who are currently on lipid-lowering pharmacological treatment in South Africa.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on lipid-lowering pharmacological treatment reaching LDL-C goals according to NCEP ATP III/Updated 2004 NCEP ATP III

SECONDARY OUTCOMES:
Proportion of patients on lipid-lowering pharmacological treatment reaching LDL-C goals according to NCEP ATP III/Updated 2004 NCEP ATP III
Proportion of patients on lipid-lowering pharmacological treatment reaching LDL-C goals according to the Fourth Joint European Task Force Guidelines/South African Guidelines in primary/secondary prevention patients, patients with metabolic syndrome
Proportion of patients on lipid-lowering pharmacological treatment reaching the non HDL-C goals according to NCEP ATP III/Updated 2004 NCEP ATP III Guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Prof F Raal, Principal Investigator — National Co-ordinator
Locations (1):
- Research Site, Johannesburg, South Africa